CLINICAL TRIAL: NCT03251183
Title: Validation of Cardiovascular Magnetic Resonance Against Invasive Haemodynamics in Patients With Heart Failure With Preserved Ejection Fraction (DECIPHER HFpEF)
Brief Title: Validation of CMR Against Invasive Haemodynamics in Patients With HFpEF
Acronym: DECIPHER-HFpEF
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Prof. Eike Nagel, Univ. Prof. Dr. med., Goethe University
Other Study IDs: Protocol_ Version 1 20170225
Record Dates: First submitted 2017-05-14; First posted 2017-08-16 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure With Normal Ejection Fraction
MeSH Terms: interventions — Blood Specimen Collection; Echocardiography; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Main group: Blood sampling Comprehensive Cardiovascular magnetic resonance (CMR) Transthoracic echocardiography (TTE) (EchoErgo) Invasive pressure-volume (PV) Loops Left ventricular (LV) biopsy
  Interventions: Diagnostic Test: Comprehensive Cardiovascular magnetic resonance (CMR); Diagnostic Test: Blood sampling; Diagnostic Test: TTE (EchoErgo); Diagnostic Test: Invasive pressure-volume (PV) Loops; Diagnostic Test: Left ventricular (LV) biopsy
- Reproducibility group: Stress-perfusion Cardiovascular magnetic resonance (CMR)
  Interventions: Diagnostic Test: Comprehensive Cardiovascular magnetic resonance (CMR); Diagnostic Test: Blood sampling
- Age/gender matched control group: Blood sampling Stress-perfusion Cardiovascular magnetic resonance (CMR) TTE (EchoErgo)
  Interventions: Diagnostic Test: Comprehensive Cardiovascular magnetic resonance (CMR); Diagnostic Test: Blood sampling; Diagnostic Test: TTE (EchoErgo)
- Healthy volunteers: Blood sampling Stress-perfusion Cardiovascular magnetic resonance (CMR) TTE (EchoErgo)
  Interventions: Diagnostic Test: Comprehensive Cardiovascular magnetic resonance (CMR); Diagnostic Test: Blood sampling; Diagnostic Test: TTE (EchoErgo)

INTERVENTIONS:
Diagnostic Test: Comprehensive Cardiovascular magnetic resonance (CMR) — Cardiovascular magnetic resonance (CMR) provides non-invasive, radiation-free and in-depth evaluation of myocardial structure and function. In addition to established tools for assessment of cardiac volume, mass, function and regional myocardial scar with late Gadolinium enhancement (LGE), several novel quantitative CMR parameters will be assessed including T1-mapping or fully quantitative perfusion Imaging.
Diagnostic Test: Blood sampling — Blood samples will eventually be analysed for markers related to heart failure (BNP/NT)-pro-BNP, myocardial inflammation and fibrosis (cytokine profiling, Galectin-3, Procollagen Type I and III, hsCRP). Whole blood will be frozen for DNA isolation and genome analysis. Peripheral blood mononuclear cells will be isolated by Ficoll in a subset of patients and will be used for RNA isolation allowing RNA-seq or reverse transcription (RT) - polymerase chain reaction (PCR) analysis.
Diagnostic Test: TTE (EchoErgo) — Measurements will include cavity dimensions, flow velocities, myocardial motion velocity and strain as well as for change of parameters during ergometric stress.
  Groups: Age/gender matched control group; Healthy volunteers; Main group
Diagnostic Test: Invasive pressure-volume (PV) Loops — Multiple parameters (including EDPVR, ESPVR, dp/dt min, Tau, Ea) will be derived from the various PV loop assessments and additional relevant parameters will be calculated. Right ventricular and pulmonary pressures including pulmonary vascular resistance will be measured with Swan-Ganz catheters using right venous femoral approach.
  Groups: Main group
Diagnostic Test: Left ventricular (LV) biopsy — A set of myocardial biopsies for each patient will be stained with Masson Trichrome for qualitative and quantitative assessment of the collagen volume fraction; fat droplets will be identified by red oil staining, Congo Red for amyloid immunohistology will be used to determine total leukocytes (CD45), T-cells (CD3) and monocytes/macrophages (CD68).
  A second set of biopsies will be frozen immediately and stored at -80°. Western blot analysis will be performed to determine alterations at the myofilament level including titin isoform composition and phosphorylation status.
  Groups: Main group

SUMMARY:
Heart failure (HF) currently affects app. 2% of the western population and app. 10% of people >75 years. In about 50% of patients with symptomatic HF ejection fraction (EF) is preserved (HF-PEF). Once patients develop symptoms, the prognosis is poor with 25% mortality at 1 year and 50% mortality at 5 years. HFpEF is one of the major unresolved areas in clinical cardiology. The diagnosis of HFpEF remains a diagnosis of exclusion and currently no non-invasive measure provides a clear diagnosis.

Cardiovascular magnetic resonance (CMR) provides non invasive and radiation free evaluation of heart structure and function. New CMR parameters offer the possibility to describe the underlying pathological and physiological changes associated with HFpEF.

The investigators propose to undertake the first systematic comparison between a CMR protocol and invasive haemodynamics as the best possible gold standard, as well as define the histopathological drivers in myocardial biopsies. The investigators will also examine the relations with tissue and serological biomarkers implicated in HFpEF and the role with standard and novel parameters by echocardiography. If successful, this study will provide tools for a reliable and accurate non-invasive characterization of patients with HFpEF, supporting the diagnosis and grading the severity of disease. This study will provide a reference basis for future diagnostic algorithms in HFpEF, both, for CMR and echocardiography, but also for their relative value in comparison to blood markers or invasive testing. In addition to a new pathway to acess the effects of current and novel therapeutic interventions, the investigators see the greatest potential in identifying a disease stage where the myocardial injury may be reversible.

ELIGIBILITY:
Main/reproducibility group:

Inclusion Criteria:

1. Ability to provide informed consent
2. Typical HF symptoms (NYHA stage II-III) within the last 6 months
3. EF > 45 % with absence of structural heart disease on echocardiography (except left ventricular hypertrophy or left atrial enlargement)
4. Echocardiographic evidence of increased left ventricular filling pressures

   1. E/E'sep >15 OR E/E'lat >12 OR Av E/E' >13 OR
   2. E/E' >9 AND left atrial (LA) volume >34 ml/m2 OR systolic pulmonary artery pressure (PAsys): >35 mmHg;
5. Indication for invasive hemodynamic work-up
6. Unclear aetiology of heart failure
7. Adults: age >18 years

Exclusion Criteria:

1. Patients unable or unwilling to provide informed consent
2. High likelihood of non-diagnostic PV loops of MR imaging (e.g. atrial fibrillation or high rate of premature ventricular contraction (PVC) (> 10 ventricular Extrasystole (VES)/minute), > 150 kg body weight, inability to lie flat or still)
3. Contraindication for invasive work-up (allergy to contrast agent, severe renal insufficiency with estimated glomerular filtration rate (eGRF) <30 ml/min)
4. Contraindications for a contrast enhanced CMR study (allergy to contrast agent, incompatible devices or implants (e.g. non-MR conditional pacemaker), severe claustrophobia)
5. Previous medical history of EF <45%
6. Imaging findings confirming a specific diagnosis of myocardial impairment (e.g. amyloid, ischaemic heart disease, valvular disease)

Age-gender matched controls:

Inclusion Criteria:

1. Ability to provide informed consent
2. No current or history of symptoms, signs or therapy for heart disease
3. EF > 45 % with absence of structural heart disease on echocardiography (except left ventricular hypertrophy or left atrial enlargement)
4. Adults: age >18 years

Exclusion Criteria:

1. Patients unable or unwilling to provide informed consent
2. High likelihood of non-diagnostic MR imaging (e.g. atrial fibrillation or high rate of PVC (> 10 VES/minute), > 150 kg body weight, inability to lie flat or still)
3. Contraindications for a contrast enhanced CMR study (allergy to contrast agent, incompatible devices or implants (e.g. non-MR conditional pacemaker), severe claustrophobia, severe renal insufficiency with eGRF <30 ml/min))
4. Previous medical history of EF <45%
5. Imaging findings confirming a specific diagnosis of myocardial impairment (e.g. amyloid, ischaemic heart disease, valvular disease)

Healthy volunteers:

Inclusion Criteria:

1. Ability to provide informed consent
2. No current or history of symptoms, signs or therapy for heart disease
3. EF ≥ 50 % with absence of structural heart disease on echocardiography

Exclusion Criteria:

1. Contraindications for an MR study
2. High likelihood of non-diagnostic MR imaging (e.g. atrial fibrillation or high rate of PVC (> 10 VES/minute), > 150 kg body weight, inability to lie flat or still)
3. Subjects unable or unwilling to provide informed consent
4. EF <50% in patient history
5. Imaging findings confirming a specific diagnosis of myocardial impairment (e.g. amyloid, ischaemic heart disease, valvular disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diagnostic criteria for HFpEF, age/gender matched controls and healty volunteers
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Significant influence of MR Imaging Parameters on a multivariate model to describe the invasive pressure volume relations (EDPVR). | up to 4 weeks. No follow up is planned.
  Using a multivariable regression analysis and a respective F test.

SECONDARY OUTCOMES:
Association between CMR T1-mapping and biopsy results. | up to 4 weeks. No follow up is planned.
  Using suitable regression and correlation Analysis.
Association between CMR flow echocardiographic flow | up to 4 weeks. No follow up is planned.
  Using suitable regression and correlation Analysis.
Association between a model for diastolic function based on CMR with a model of diastolic function based on echocardiography | up to 4 weeks. No follow up is planned.
  Using suitable regression and correlation Analysis.
Association between CMR function and echocardiographic function | up to 4 weeks. No follow up is planned.
  Using suitable regression and correlation Analysis.
Discriminatory capacity of a multivariate model of invasive and a multivariate model of non-invasive variables. | up to 4 weeks. No follow up is planned.
  Using the patient and control groups with comparative ROC analysis and DeLong tests.
Reproducibility at one site. | up to 4 weeks. No follow up is planned.
  Using respective intra-class correlations in the groups with multiple measurements.
Variability between the different sites. | up to 4 weeks. No follow up is planned.
  Using respective intra-class correlations in the groups with multiple measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Eike C Nagel, MD, PhD, Principal Investigator — Goethe University Frankfurt
Locations (7):
- Germany (7):
  - University Hospital Frankfurt, Frankfurt am Main, Hesse
  - Kerckhoff Klinik, Bad Nauheim
  - Charite Centrum Herz-, Kreislauf- und Gefäßmedizin, Berlin
  - University Hospital Göttingen, Göttingen
  - University Hospital, Heidelberg
  - Herzzentrum Leipzig, Leipzig
  - Uniersity Hospital Mainz, Mainz

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared with other researchers within the German Centre for Cardiovascular Research (DZHK) via the Use and Access Rules
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: 1 year after finalization of primary analysis
Access Criteria: Via Use and Access Policy of DZHK
URL: https://www.dzhk.de